CLINICAL TRIAL: NCT01533610
Title: The Efficacy of Stellate Ganglion Block as PTSD Therapy: A Pilot Study
Brief Title: The Efficacy of Stellate Ganglion Block as Post-traumatic Stress Disorder (PTSD) Therapy: A Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: #1125
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress disorder; Stellate ganglion; cervical plexus; local anesthesia; anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Cervical Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stellate ganglion block — Local anesthesia applied to the stellate ganglion in the neck
  Other Names: Cervical plexus block

SUMMARY:
RATIONALE: A stellate ganglion nerve block may help relieve symptoms of post-traumatic stress disorder (PTSD).

PURPOSE: This pilot clinical trial is studying the efficacy of a stellate ganglion nerve block in veterans to reduce the symptoms of PTSD in relatively long-standing (Vietnam era) induced or relatively recently induced PTSD (from deployment in Afghanistan or Iraq as part of Operations Enduring Freedom (OEF), Iraqi Freedom (OIF), and New Dawn (OND).

DETAILED DESCRIPTION:
Objectives:

1. Stellate ganglion blocks will be performed in a small sample (n = 12) of the local patient population that suffers from PTSD in order to replicate other preliminary findings.
2. The parameters that lead to a successful treatment response will be evaluated by comparing and contrasting the results obtained in younger (n=6) OEF/OIF generation veterans versus older (n=6) Vietnam generation veterans.
3. The individual difference variables that might lead to successful treatment responses will be studied by obtaining correlative measures of psychological and psychometric data and responses to standardized tests.

Research Design:

This is an open label unblinded clinical pilot case series study to determine the efficacy of stellate ganglion blockade for relief of PTSD symptoms in the Long Beach VA healthcare population.

ELIGIBILITY:
Inclusion Criteria:

* Include significant PTSD symptoms with severe hyper-arousal symptoms.
* Clinician Administered PTSD Scales (CAPS) score, with a total score ≥ 50 needed for enrollment.
* Hyper-arousal severity identified by a high score on the CAPS D scale and a ≥ 10 beat per minute increase in heart rate during the subject's verbal recollection of a standardized version of their traumatic exposure.

Exclusion Criteria:

* Include psychiatric and medical conditions that would make patients poor candidates for an outpatient procedure.
* Subjects must be able to be cooperative for the procedure and free of significant medical problems that would pose a constant threat to life.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Difference in CAPS score activity | Baseline and weeks 1, 4, 12 and 26

SECONDARY OUTCOMES:
Depression scale | Baseline and weeks 1, 4, 12 and 26
Anxiety scale | Baseline and weeks 1, 4, 12 and 26
Quality of life scale | Baseline and weeks 1, 4, 12 and 26
Biophysical responses | Baseline and weeks 1, 4, 12 and 26

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Alkire, MD, Principal Investigator — Long Beach VA Healthcare system
Locations (1):
- VA Long Beach Healthcare system, Long Beach, California, United States